CLINICAL TRIAL: NCT00052182
Title: A Single Center Phase I Safety and Immunogenicity Study of Epimmune HIV-1 CTL Epitope-Based DNA Vaccine (EP HIV-1090) for Immunotherapy of HIV-1 Infected Individuals Receiving Highly Active Antiretroviral Therapy (HAART)
Brief Title: Safety of and Immune System Response to an HIV Vaccine (EP HIV-1090) in HIV Infected Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: P01AI048238-03 (NIH); IPCP 01
Record Dates: First submitted 2003-01-24; First posted 2003-01-27 (Estimated); Last update posted 2007-10-23 (Estimated); Status verified 2007-09

CONDITIONS: HIV Infections
Keywords: HIV Therapeutic Vaccine; CTL Epitope; Treatment Experienced
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- 1 (Experimental): Immunization on Day 0 and Weeks 4, 8, and 16
  Interventions: Biological: EP HIV-1090

INTERVENTIONS:
Biological: EP HIV-1090

SUMMARY:
HIV-1-infected patients who have been treated with anti-HIV drugs for a long time may have weakened immune responses to HIV. The DNA-based vaccine in this study is designed to boost the immune system's responses against many HIV-1 proteins. The main purposes of this study are to test the safety of this HIV vaccine (EP HIV-1090) and to test whether the vaccine can stimulate immune system responses in people who have HIV-1 infection.

DETAILED DESCRIPTION:
Significant data support the hypothesis that HIV-specific cytotoxic T lymphocyte (CTL) responses contribute to the control and potential clearance of the virus. Vaccines designed specifically to induce CTL responses are likely to be well suited for treatment of HIV infection. The conceptual basis of the EP HIV-1090 vaccine is the use of highly defined CTL epitopes as the vaccine immunogen. The vaccine is formulated with a water-soluble polymer that stabilizes and protects the DNA and facilitates uptake by cells. Preclinical studies have shown that the vaccine induces strong CTL responses in animal models. This study will evaluate the safety and tolerability of the vaccine and the immune response to the vaccine in HIV-1-infected individuals who are being treated with highly active antiretroviral therapy (HAART) and have a CD4 count of 350 cells/mm3 or more and fully suppressed viral replication on stable HAART.

Each patient will receive a total of four immunizations to be given at Day 0 and at Weeks 4, 8, and 16. Participants will be randomly assigned to receive either vaccine or placebo. Ten patients will be assigned to each dose group; eight will receive active vaccine and two will receive placebo. The injections will be delivered intramuscularly into the deltoid muscle. In addition to undergoing standard safety exams, patients will have blood drawn for use in evaluating the immunogenicity of the vaccine. The treatment duration will be 16 weeks and patient will be followed for safety and immune responses for an additional 24 weeks after they complete vaccination; the total study is estimated to take 18 months.

ELIGIBILITY:
Inclusion Criteria

* Documented HIV-1 infection
* Taking HAART for 6 months or longer and on stable HAART for at least 4 weeks
* Plasma HIV-1 viral load of less than 400 copies/ml for at least 6 months prior to study entry
* CD4 count of 350 cells/mm3 or more within 30 days of entry

Exclusion Criteria

* Immunomodulatory agents
* Prior receipt of experimental HIV vaccines in the 5 years prior to study entry
* Hepatitis B surface antigen or hepatitis C virus antibody positive

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2002-10

PRIMARY OUTCOMES:
Safety and efficacy of four intramuscular doses of EP HIV-1090 to HIV infected participants using highly active antiretroviral therapy (HAART), who have a viral load less than 400 | Throughout study

SECONDARY OUTCOMES:
Peripheral blood CD8 T-cell (CTL) responses to vaccine, compared to placebo | Throughout study
CD4 T-cell count and viral load in patients continuing HAART following vaccination or receipt of placebo | Throughout study
Clinical signs and symptoms and development of AIDS-defining clinical events following vaccination or receipt of placebo in participants who remain on HAART | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Constance Benson, MD, Study Chair — University of California, San Diego
Locations (1):
- University of Colorado, Health Science Center, Denver, Colorado, United States

REFERENCES:
- [Background] Wilson CC, McKinney D, Anders M, MaWhinney S, Forster J, Crimi C, Southwood S, Sette A, Chesnut R, Newman MJ, Livingston BD. Development of a DNA vaccine designed to induce cytotoxic T lymphocyte responses to multiple conserved epitopes in HIV-1. J Immunol. 2003 Nov 15;171(10):5611-23. doi: 10.4049/jimmunol.171.10.5611. PMID 14607970